CLINICAL TRIAL: NCT04879654
Title: Phase II, Single-arm, Prospective Clinical Study of Toripalimab Combined With Radiotherapy and Chemotherapy in the Treatment of Sinonasal Malignant Mucosal Melanoma（SNMM） After Endoscopic Surgery
Brief Title: Toripalimab Combined With Radiotherapy and Chemotherapy in the Treatment of SNMM After Endoscopic Surgery
Acronym: SNMM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Hongmeng Yu, MD,PhD, Eye & ENT Hospital of Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNMM-SA-V1
Record Dates: First submitted 2021-05-05; First posted 2021-05-10 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Malignant Melanoma; Sinonasal Melanoma
MeSH Terms: conditions — Melanoma | interventions — Endoscopy; Radiotherapy; Drug Therapy; toripalimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- endonasal endoscopic surgery with adjuvant therapy (Experimental): endonasal endoscopic surgery followed by Toripalimab,radiotherapy and/or chemotherapy
  Interventions: Procedure: endoscopic surgery

INTERVENTIONS:
Procedure: endoscopic surgery — endoscopic surgery followed by multimodality treatment including radiotherapy,Toripalimab,and/or chemotherapy
  Other Names: radiotherapy; chemotherapy; Toripalimab

SUMMARY:
Phase II, single-arm, prospective clinical study of Toripalimab(a PD-1 antibody) combined with radiotherapy and chemotherapy in the treatment of sinonasal malignant mucosal melanoma after endoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

1.Pathologically diagnosed as sinonasal malignant mucosal melanoma, locally resectable and no contraindication for surgery or radiation. 2.T3 and T4. 3.Age ≥18 year-old 4.No distant metastasis 5.No head and neck radiation and systemic anti-tumor therapy performed in the past 5 years. 6.The performance status of the Eastern Cooperative Oncology Group(ECOG) is 0-2 points and surgery after general anesthesia and postoperative radiation could be tolerated. 7.Accepted organ function

Exclusion Criteria:

1. Patients who refused to sign informed consent. 2. Have received radioactive seed implantation in the treatment area. 3. Suffer from uncontrolled disease which could interfere treatment. 4. Suffered from another malignant tumor or multiple primary tumors at the same time within 5 years (excluding fully treated basal cell or squamous cell skin cancer, cervical cancer in situ, etc.). 5. The patient has surgical contraindications: such as severe cardiopulmonary disease, coagulation dysfunction and so on. 6.The patients have autoimmune diseases. 7. The patient is using immunosuppressive agents or systemic hormone therapy to achieve the purpose of immunosuppression (dose>10mg/day prednisone or other curative hormones), and continues to use it within 2 weeks before the first administration; 8. Severe allergic reaction to other monoclonal antibodies; 9. Previously received PD-1 monoclonal antibody, CTLA-4 monoclonal antibody (or any other antibody that acts on T cell co-stimulation or checkpoint pathway) treatment; 10. Live vaccines have been inoculated within 4 weeks before the first administration or during the study period; 11. The patient has any situation that may hinder study compliance or the safety during the study period.12. Existence of serious neurological or psychiatric diseases, such as dementia and seizures; 13. Uncontrolled active infection. 14. Pregnant or breastfeeding women. 15. Those who have no personal freedom and independent capacity for civil conduct;p. 16. There are other situations that are not suitable for entry into the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From date of first treatment until the date of death from any cause,through study completion,up to 3 years.]
  3 year Overall Survival rate

SECONDARY OUTCOMES:
progression free survival | From date of first treatment until the date of first documented progression or date of death from any cause, whichever came first，through study completion,up to 3 years.
  the date of first treatment to the first recording of disease progression or death from any cause.

OTHER OUTCOMES:
Local progression free survival | From date of first treatment to local failure or date of death from any cause,through study completion,up to 3 years.
  the date of first treatment to local failure or death
Regional progression free survival | From date of first treatment to regional failure or date of death from any cause, through study completion,up to 3 years.
  the date of first treatment to regional failure or death
Distant metastasis free survival | From date of first treatment to distant metastasis or date of death from any cause, through study completion,up to 3 years.]
  the date of first treatment to distant metastasis or death
Toxicities | From date of first treatment through study completion,up to 3 years.
  Using CTCAE Version5.0 to evaluate

CONTACTS AND LOCATIONS:
Overall Officials: Hongmeng Yu, MD,PHD, Principal Investigator — Eye&ENT Hospital,Fudan University
Locations (1):
- Eye& ENT Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes